CLINICAL TRIAL: NCT05660395
Title: A Phase 1b Open-Label Study to Evaluate the Pharmacokinetics and Safety of Loncastuximab Tesirine in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma or High-grade B-cell Lymphoma With Hepatic Impairment (LOTIS-10)
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Loncastuximab Tesirine in Participants With Relapsed or Refractory Diffuse Large B-cell Lymphoma or High-grade B-cell Lymphoma With Hepatic Impairment (LOTIS-10)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ADCT-402-107; 2021-005209-29 (EudraCT Number)
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B-Cell Lymphoma; High-grade B-cell Lymphoma
Keywords: Loncastuximab Tesirine; Lymphoma; DLBCL; HGBCL; Hepatic Impairment
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Normal Hepatic Function (Experimental): Participants will receive loncastuximab tesirine 0.15 mg/kg once every 3 weeks (Q3W) for two cycles, then 0.075 mg/kg Q3W for subsequent cycles (1 cycle = 21 days).
  Participants who have a toxicity meeting the criteria for dose reduction will have subsequent doses reduced by 50%. If the toxicity recurs, subsequent doses must be reduced by an additional 50%. A maximum of 2 dose reductions are allowed. Participants who have a toxicity meeting the criteria for dose reduction following Cycle 2 will receive the protocol-specified dose of 50% of initiate dose for Cycle 3, i.e., they will not have an additional dose reduction for Cycle 3.
  Interventions: Drug: Loncastuximab Tesirine
- Arm B: Moderate Hepatic Impairment (Experimental): Participants will receive loncastuximab tesirine in a standard 3+3 dose-escalation design. Initial dose will be 0.09 mg/kg Q3W for two cycles, then 0.045 mg/kg Q3W for subsequent cycles (1 cycle = 21 days). The highest dose possibly administered will be 0.15 mg/kg Q3W.
  Participants who have a toxicity meeting the criteria for dose reduction will have subsequent doses reduced by 50%. If the toxicity recurs, subsequent doses must be reduced by an additional 50%. A maximum of 2 dose reductions are allowed. Participants who have a toxicity meeting the criteria for dose reduction following Cycle 2 will receive the protocol-specified dose of 50% of initiate dose for Cycle 3, i.e., they will not have an additional dose reduction for Cycle 3.
  Interventions: Drug: Loncastuximab Tesirine
- Arm C: Severe Hepatic Impairment (Experimental): Participants will receive loncastuximab tesirine in a standard 3+3 dose-escalation design. Initial dose will be 0.09 mg/kg Q3W for two cycles, then 0.045 mg/kg Q3W for subsequent cycles (1 cycle = 21 days). The highest dose possibly administered will be 0.15 mg/kg Q3W.
  Participants who have a toxicity meeting the criteria for dose reduction will have subsequent doses reduced by 50%. If the toxicity recurs, subsequent doses must be reduced by an additional 50%. A maximum of 2 dose reductions are allowed. Participants who have a toxicity meeting the criteria for dose reduction following Cycle 2 will receive the protocol-specified dose of 50% of initiate dose for Cycle 3, i.e., they will not have an additional dose reduction for Cycle 3.
  Interventions: Drug: Loncastuximab Tesirine

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Intravenous (IV) Infusion
  Other Names: Zynlonta; ADCT-402

SUMMARY:
The primary objective of this study is to determine the recommended dosing regimen of loncastuximab tesirine in diffuse large B-cell lymphoma (DLBCL) or high-grade B-cell lymphoma (HGBCL) participants with moderate and severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or older
* Pathologic diagnosis of relapsed (disease that has recurred following a response) or refractory (disease that failed to respond to prior therapy) DLBCL not otherwise specified, DLBCL arising from low grade lymphoma, and high-grade B-cell lymphoma (2016 World Health Organization classification) who have received at least one systemic treatment regimen
* Measurable disease as defined by the 2014 Lugano Classification
* Normal hepatic function or hepatic impairment as defined by the National Cancer Institute Organ Dysfunction Working Group hepatic impairment classification:

  * Arm A Normal hepatic function: bilirubin and aspartate aminotransferase (AST) ≤ upper limit of normal (ULN)
  * Arm B Moderate hepatic impairment: bilirubin > 1.5 × to 3 × ULN (any AST)
  * Arm C Severe hepatic impairment: bilirubin > 3 × ULN (any AST)
* ECOG performance status 0 to 2 for participants with normal hepatic function. ECOG 0 to 3 for participants with moderate or severe hepatic impairment
* Adequate organ function
* Women of childbearing potential (WOCBP)* must agree to use a highly effective method of contraception from the time of giving informed consent until at least 10 months after the last dose of study drug. Men with female partners who are of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of the first dose until at least 7 months after the last dose of study drug.

Exclusion Criteria:

* Previous therapy with loncastuximab tesirine
* Allogenic or autologous stem cell transplant within 60 days prior to start of study drug (C1D1)
* Human immunodeficiency virus (HIV) seropositive
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis
* Lymphoma with active central nervous system involvement at the time of screening, including leptomeningeal disease
* Breastfeeding or pregnant
* Significant medical comorbidities
* Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy, within 14 days prior to start of study drug (C1D1), except shorter if approved by the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Moderate or Severe Hepatic Impairment Who Experience a Dose-Limiting Toxicity (DLT) | Day 1 to Day 21 of Cycle 1, where a cycle is 21 days

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Time to Cmax (Tmax) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Area Under the Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Area Under the Concentration-time Curve from Time Zero to the End of the Dosing Interval (AUCtau) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Area Under the Concentration-time Curve from Time Zero to Infinity (AUCinf) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Apparent Terminal Elimination Half-life (Thalf) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Apparent Clearance (CL) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Apparent Steady-state Volume of Distribution (Vss) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Accumulation Index (AI) of Loncastuximab Tesirine and SG3199 in Serum | Day 1 up to 1 year
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 3 years
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Up to approximately 1 year
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Delay | Up to approximately 1 year
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Interruption | Up to approximately 1 year
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Reduction | Up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in Safety Laboratory Values | Baseline up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in Vital Signs | Baseline up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in 12-Lead Electrocardiogram (ECG) Measurements | Baseline up to approximately 1 year
Overall Response Rate (ORR) | Up to approximately 3 years
Duration of Response (DOR) | Up to approximately 3 years
Complete Response (CR) Rate | Up to approximately 3 years
Progression-Free Survival (PFS) | Up to approximately 3 years
Relapse-Free Survival (RFS) | Up to approximately 3 years
Overall Survival (OS) | Up to approximately 3 years
Number of Participants With Anti-drug Antibody (ADA) Titers to Loncastuximab Tesirine | Day 1 up to 1 year

CONTACTS AND LOCATIONS:
Locations (14):
- The Oncology Institute of Hope & Innovation - Lynwood, Lynwood, California, United States
- Brazil (6):
  - Hospital Sírio-Libanês - Brasília, Brasília
  - Hospital Mãe de Deus - Centro Integrado de Oncologia, Porto Alegre
  - Hospital Sírio-Libanês - São Paulo, São Paulo
  - A Beneficência Portuguesa de São Paulo - Unidade Mirant, São Paulo
  - Hospital 9 de Julho, São Paulo
  - Albert Einstein Israelite Hospital, São Paulo
- South Korea (5):
  - Kyungpook National University Chilgok Hospital, Daegu, Daegu Gwang'yeogsi
  - Dong-A University Hospital, Pusan, Gyeongsangnam-do
  - Korea University Anam Hospital, Seoul, Seongbuk District
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Severance Hospital, Seoul, Seoul Teugbyeolsi
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: No